CLINICAL TRIAL: NCT06359119
Title: Implementation of Apnoea Test for Patients With Suspected Brain Death (IMAPing SUBDEP)
Brief Title: Implementation of Apnoea Test for Patients With Suspected Brain Death
Status: Not yet recruiting | Type: Observational
Sponsor: Kiskunhalas Semmelweis Hospital the Teaching Hospital of the University of Szeged (Other Government)
Collaborators: Veszprém County Ferenc Csolnoky Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: IMAPing SUBDEP
Record Dates: First submitted 2024-03-27; First posted 2024-04-11 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Brain Death
Keywords: brain death determination; apnoea test; survey
MeSH Terms: conditions — Brain Death

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study consists of a survey created for intensive care physicians regarding their current practice of the implementation of apnoea test for patients with suspected brain death.

DETAILED DESCRIPTION:
Although the apnoea test is part of nearly all protocols for determining brain death; implementation significantly differs among intensive care physicians according to national-level acts, national society protocols or local protocols.

This cross-sectional study is based on an international, web-based questionnaire created for intensive care physicians, consisting of 25 questions in English.

The survey will provide a current state of the practice of apnoea testing in patients with suspected brain death. The results can support the determination of future acts to standardize the apnoea test process.

The given answers are anonymous. The e-mail address of the respondent is not recorded. Answers are treated solely for scientific purposes.

ELIGIBILITY:
Inclusion Criteria:

* Physicians working in intensive care units

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any physician working in intensive care can fill the form and participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of apnoea tests | last 1 year
  How much apnoea test is required for brain death determination.
Timeframe between apnoea tests | last 1 year
  If more than 1 apnoeae test is reuired for brain death determination, how many hours should elapse between the two tests.
Preoxygenation | last 1 year
  For how long (in minutes) the patient is preoxygenated before the apnoea test.
Baseline arterial carbon dioxide (CO2) level | Last 1 year
  What is the required arterial partial CO2 pressure (PaCO2) before apnoea testing, confirmed by arterial blood gas measurement?

SECONDARY OUTCOMES:
Detection of possible spontaneous breath movements | last 1 year
  To determine if any observation method other than visualisation by the observer is used to determine possible spontaneous breath movements during the apnoea test.
Satisfaction with current practice | last 1 year
  Surveying the satisfaction of physicians with current practice regarding the method of the detection of spontaneous breath movements on a 4 grade scale (1 - non-reliable to 4 - very reliable).

OTHER OUTCOMES:
Continuous positive airway pressure (CPAP) | last 1 year
  If a CPAP system is used during apnoea test, what is the value of positive end-expiratory pressure (PEEP) in H2Ocm.